CLINICAL TRIAL: NCT04257604
Title: A Multicenter, Prospective, Real-life Observational Study of Perampanel as Add-on Therapy in Adult and Adolescent Patients With Focal Seizures (A Mirroring Clinical Practice Study of Perampanel in Adults and Adolescents) (The AMPA Study)
Brief Title: A Study of Perampanel as Add-on Therapy in Adult and Adolescent Participants With Focal Seizures
Status: Completed | Type: Observational
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E2007-M044-501
Record Dates: First submitted 2020-01-10; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-01

CONDITIONS: Partial Seizures
Keywords: Perampanel; Partial seizures; Focal seizures
MeSH Terms: conditions — Seizures | interventions — perampanel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perampanel: Participants with partial-onset seizures, with or without secondary generalization will receive perampanel tablets as add-on therapy according to the approved summary of product characteristics (SmPC) after the baseline visit as part of the clinical practice and will be observed after 3 months (visit 1), 6 months (visit 2), and 12 months (final visit).
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — Perampanel tablets.
  Other Names: Fycompa; E2007

SUMMARY:
The primary objective of the present study will be to assess the effectiveness of add-on perampanel in participants with focal seizures in a real-life clinical setting.

ELIGIBILITY:
Inclusion Criteria:

1. Prescribe perampanel according to the approved indication
2. Participants with focal seizures with or without secondary generalization
3. Participants with seizure frequency data available at the baseline visit
4. Based on the physician's clinical judgment, the participant seizure activity is not controlled sufficiently with the current treatment with 1-3 AEDs and it is in the participants best interest to be prescribed adjunctive perampanel
5. The decision to prescribe perampanel is made by the physician before and independently of his/her decision to include the participant in the study
6. Treatment with perampanel is not yet started before baseline

Exclusion Criteria:

1. Participants contraindicated for perampanel use (according to SmPC)
2. Participants with moderate to severe renal impairment
3. Participants with severe hepatic impairment
4. Pregnant or lactating women
5. Participants suffering from clinically significant psychiatric illness, psychological or behavioral problems which could interfere with study participation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with epilepsy aged 12 years or older.
Sampling Method: Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2016-01-03 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage Change From Baseline in all Seizures Frequency at Month 6 | Baseline, Month 6
  Seizure frequency is derived from information (seizure count and type) recorded in participant diary. Seizure frequency is based on the number of seizures per 28 days, calculated as the number of seizures over the entire time interval divided by the number of days in the interval and multiplied by 28.

SECONDARY OUTCOMES:
Percentage of Participants Remaining on Perampanel at Months 6 and 12 | Months 6 and 12
  The retention rate is defined as the percentage of participants remaining on perampanel, starting from the first dose of study drug.
Percentage of Participants With Adverse Drug Reactions (ADRs) and Serious Adverse Drug Reactions (SADRs) | Up to Month 12
  ADR is a noxious and unintended response to a medicinal product related to any dose. A causal relationship between the medicinal product and the adverse response is at least a reasonable possibility. A SADR is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization¸ results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Percentage of Participants Who Withdraw due to ADR | Up to Month 12
  ADR is a noxious and unintended response to a medicinal product related to any dose. A causal relationship between the medicinal product and the adverse response is at least a reasonable possibility.
Percentage of Participants Who Withdraw due to Lack of Efficacy | Up to Month 12
  Lack of efficacy is if the participant had poor seizure control (defined as experiencing a seizure despite being on the maximum dose for equal to 2 weeks). The participant can withdraw at any time due to lack of efficacy.
Mean Change From Baseline in the Number of Concomitant Anti-epileptic Drugs (AEDs) | Baseline up to Month 12
  Change from baseline in the number of concomitant AEDs along with the Perampanel will be reported.
Percentage of Participants With at Least 50 Percent (%) and 75% Reduction From Baseline in All Seizure Frequency at Months 3, 6 and 12 | Baseline, Months 3, 6, and 12
  A 50% or 75% responder rate is percentage of participants who experience at least 50% or 75% reduction in all seizure frequency during the study.
Percentage of Participants With at Least 50% and 75% Reduction From Baseline in Secondarily Generalized Tonic-clonic Seizures (SGTCS) Frequency at Months 3, 6 and 12 | Baseline, Months 3, 6, and 12
  A 50% or 75% responder rate for SGTCS is percentage of participants who experience at least 50% or 75% reduction of SGTCS frequency during the study. Focal to bilateral toni-clonic seizures (FBTCS) replaces older term SGTCS. FBTCS is a seizure type with focal onset, with awareness or impaired awareness, either motor or nonmotor, progressing to bilateral tonic-clonic activity.
Percentage of Participants Who Were Seizure-free | Up to Month 12
  Participants will be considered seizure-free if participants will not experience any partial-onset seizure during the study.
Median Percentage Change From Baseline in All Seizure Frequency at Months 3 and 12 | Baseline, Months 3 and 12
  Seizure frequency is based on the number of seizures per 28 days, calculated as the number of seizures over the entire time interval divided by the number of days in the interval and multiplied by 28.
Median Percentage Change From Baseline in SGTCS Frequency at Months 3, 6 and 12 | Baseline, Months 3, 6, and 12
  SGTCS frequency is based on the number of SGTC seizures per 28 days, calculated as the number of SGTC seizures over the entire time interval divided by the number of days in the interval and multiplied by 28. FBTCS replaces older term SGTCS. FBTCS is a seizure type with focal onset, with awareness or impaired awareness, either motor or nonmotor, progressing to bilateral tonic-clonic activity.
Mean Change From Baseline in 31-item Quality of Life in Epilepsy (QOLIE-31) Questionnaire Score in Adult Participants at Month 6 and 12 | Baseline, Months 6 and 12
  The Italian version of the QOLIE-31 will be used in this study. The QOLIE-31 inventory is a 31-item self-administered questionnaire evaluating Quality of Life (QOL) perception in adults 18 years or older with epilepsy in 7 domains: seizure worry, emotional wellbeing, energy/fatigue, cognitive functioning, medication effects, social functioning, overall QOL. The overall score is derived by weighing and then summing the 7 domain scores. Pre-coded numeric values for some domains are such that a higher number reflects a more favorable health state; others are such that a higher number reflects a less favorable state. Pre-coded values are converted to 0 to 100 point scores; a higher converted score indicates a higher self-reported QOL.
Mean Change From Baseline in Epworth Sleepiness Scale (ESS) Score in Adult Participants at Months 3, 6, and 12 | Baseline, Months 3, 6, and 12
  The ESS is a self-administered questionnaire with 8 questions. It provides a measure of a participant's general level of daytime sleepiness, or average sleep propensity in daily life. The ESS asks the participant to rate, on a 4-point scale (0 [low] to 3 [high]) his or her usual chances of dozing off or falling asleep in 8 different situations or activities that most people engage in as part of their daily lives. The total ESS score provides an estimate of a general characteristic of each person's average level of sleepiness in daily life (0= no chance of dozing/no daytime sleepiness to 24=high chance of dozing/lots of daytime sleepiness).
Mean Change From Baseline in Irritability With Epilepsy Questionnaire Score (I-Epi) in Adult Participants at Months 3, 6, and 12 | Baseline, Months 3, 6, and 12
  I-Epi is a questionnaire specific for the assessment of irritability in adult participants with epilepsy. I-Epi is an 18-item self-administered questionnaire based on four dimensions related to irritability in participants affected by epilepsy (physical functioning, verbal functioning, temperamental functioning, and epilepsy functioning). Participants have to rate their irritability level on a 6-point Likert scale where 1="never," 2="almost never," 3="rarely,"4="sometimes," 5="often," and 6="always". Higher score means more irritability.
Regression Coefficient For Predictive Factors in Response to Perampanel | Up to Month 12
  Predictive factors include age, age greater than or equal to (>=) 60 years, age less than (<) 18 years, gender, body mass index (BMI), age at seizure onset, age at diagnosis of epilepsy, time since diagnosis of epilepsy, baseline 28-day seizure frequency, seizure type, epilepsy familiarity (yes or no), epilepsy surgery (yes or no), focal known etiology (yes or unknown), number of seizures at baseline, number of AEDs at baseline, presence or absence of enzyme-inducing AEDs, eziologia vascolare (yes versus other). Regression coefficient will be determined to characterize the association between predictive factors and response to perampanel.

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.